CLINICAL TRIAL: NCT07336173
Title: Role of Uterine Artery Doppler Indices and Sonographic Measurement of Uterocervical Angle in Predicting Preterm Labor
Brief Title: Uterine Artery Doppler Indices and Uterocervical Angle Measurment in Prediction of Preterm Labor
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nourhan Moustafa Elsayed Shalaby, Resident physician doctor, Kafrelsheikh University
Other Study IDs: KFSIRB200-597
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Trans abdominal ultrasound will be used to measure uterine artery doppler indices Trans vaginal ultrasound will be used to measure anterior uterocervical angle

SUMMARY:
The goal of this observational study is to evaluate the role of uterine artery doppler indices and uterocervical angle measurement in prediction of preterm labor .The main question it aims to answer is:

Does combination of both uterine artery doppler indices and uterocervical angle measurement increase sensitivity and specificity for prediction of established preterm labor ? Participants already performing uterine artery doppler as part of their regular antenatal care .measurement of anterior uterocervical angle will be added between 24 to 34 weeks gestation to predict preterm labor in candidates .

DETAILED DESCRIPTION:
In this study the aim is to evaluate the combined predictive value of both uterine artery doppler and uterocervical angle measurement in a prospective cohort study design to predict preterm labor . The abnormal mid-trimester uterine artery resistance, pulsatility index and diastolic notching measured with Doppler sonography is known to be predictive for preeclampsia and, hence, for iatrogenic Preterm labor. It will be measured via trans abdominal approach.

The measurement of UCA in the second trimester of pregnancy is strongly associated with the occurrence of spontaneous Preterm labor and will be measured via transvaginal approach .

Both measurement will be conducted between 24 to 34 weeks gestational .

ELIGIBILITY:
Inclusion Criteria:

1. Patient who will give verbal & written will informed consent.
2. Pregnant women between 18 and 40 years old of age
3. Singleton pregnancy
4. Gestational age will be confirmed by first trimester ultrasound scan (<14 weeks).
5. Gestational age between 24 and 34 weeks .
6. Threatened preterm labor which is defined as:

Presence of at least one uterine contraction every 10 minutes lasting ≥30 seconds . Cervical dilatation ≤3 cm . Cervical effacement <80%.

Exclusion Criteria:

Obstetric:

1. Ruptured membranes
2. Clinical evidence of Chorioamnionitis.
3. Fetal compromise on evaluation.
4. Severe obstetric complications (e.g., severe Preeclampsia, Eclampsia).
5. Diagnosed intrauterine growth restriction (IUGR).
6. Congenital fetal anomalies.
7. Multiple pregnancies.
8. Prior cervical surgery (e.g., cone biopsy, cerclage).

Non-Obstetric:

1. Significant maternal medical disorders (e.g., chronic hypertension, diabetes mellitus, liver dysfunction).
2. Severe non-obstetric complications (e.g., acute abdomen).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant females
Study Population: Eligible participants will be recruited among those attending the antenatal clinic or Obstetrics Emergency Unite at Kafrelsheikh University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy performance of uterine artery Doppler indices and uterocervical angle assed by ultrasound for prediction of preterm labor | From 24 to 34 weeks gestation
  Its hypothesized that:
  Abnormal uterine artery Doppler indices and an abnormal (acute) uterocervical angle (< 95°) are significant predictors of preterm labor. The combination of these two parameters will enhance the sensitivity and specificity of preterm labor prediction.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr elsheikh university hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No